CLINICAL TRIAL: NCT04672187
Title: Middle Ear Status in Cholesteatoma: the Associations of Preoperative Computed Tomography Scans, Audiologic Assessment, and Intraoperative Endoscopic Findings
Brief Title: Associations of Pre- and Intraoperative Endoscopic Findings of Middle Ear Status in Cholesteatoma
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Yuvatiya Plodpai, Associate professor, Prince of Songkla University
Other Study IDs: EC-60-237-131
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Middle Ear Cholesteatoma
Keywords: endoscopic,cholesteatoma,audiogram, air-bone gap
MeSH Terms: conditions — Cholesteatoma, Middle Ear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the accuracy of preoperative HRCT of the temporal bone combined with the preoperative audiologic assessment compared with the intraoperative endoscopic middle ear finding.

DETAILED DESCRIPTION:
The information of the preoperative HRCT scanning of the middle ear cavity in cholesteatoma combined with the preoperative audiologic assessment could be informed the intraoperative middle ear finding in the patients who were diagnosed with chronic otitis media with cholesteatoma, which influence the plan of surgical management. Whether these preoperative assessments can predict the intraoperative finding is unclear. The aim of this study is to assess the accuracy of preoperative HRCT of the temporal bone combined with the preoperative audiologic assessment compared with the intraoperative endoscopic middle ear finding.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study had otorrhea, hearing loss, or aural fullness that last more than 3 months. Otological examination revealed tympanic membrane perforation or retraction, along with cholesteatoma.

Exclusion Criteria:

* Patients who had a previous temporal bone fracture, concomitant with congenital craniofacial anomalies, or underwent previous otologic surgery were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We prospectively evaluated the preoperative HRCT scanning of the temporal bone and preoperative audiologic assessment compared with an intraoperative endoscopic finding of patients who were diagnosed with chronic otitis media with cholesteatoma and scheduled to a primary surgery at Otolaryngology department, Songklanagarind hospital, Prince of Songkla University between November 2017 to November 2019.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
predictive factor of intraoperative endoscopic finding from preoperative ct finding and preoperative audiological assessment | 2 years
  the association of preoperative ct finding and preoperative audiological assessment compared with intraoperative endoscopic middle ear finding in middle cholestaetoma

SECONDARY OUTCOMES:
accuracy between preoperative ct finding and intraoperative endoscopic finding | 2 years
  accuracy between preoperative ct finding and intraoperative endoscopic finding of middle ear cholesteatoma

CONTACTS AND LOCATIONS:
Overall Officials: Yuvatiya Plodpai, MD, Principal Investigator — Faculty of Medicine, Prince of Songkla University
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand